CLINICAL TRIAL: NCT01868204
Title: Pharmacogenetic Study of Neurofunctional Brain Areas Related to Food Craving in Obese Patients With Binge Eating Disorder Treated With Topiramate
Brief Title: Pharmacogenetic and Neurofunctional Brain Areas Study in Obese Patients With Binge Eating Disorder
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Instituto Nacional de Psiquiatría Dr. Ramón de la Fuente (Other)
Responsible Party: Principal Investigator, Beatriz Elena Camarena Medellin, Medical Science Investigator, Instituto Nacional de Psiquiatría Dr. Ramón de la Fuente
Other Study IDs: TOPMATOBE3002; IC092024.0 (Other: IC092024.0)
Record Dates: First submitted 2013-05-30; First posted 2013-06-04 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-05

CONDITIONS: Obesity; Binge Eating Disorder
Keywords: Obesity; Binge eating disorder; Pharmacogenetic; Food craving; Brain areas; Topiramate
MeSH Terms: conditions — Obesity; Binge-Eating Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Genomic DNA will be extracted from 5 ml of peripheral blood using standard method.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Adoption, twin and family studies have reported that obesity has a strong heritable component and in particular, it has been suggested that BMI in adults is due to genetic influence rather than shared family environment. Binge eating in obese patients was described. Therefore, it has been proposed that binge eating disorder (BED) may contribute to obesity in some individuals.

Pharmacological studies reported that topiramate plays an important role in the treatment of binge eating disorder. It has been observed improvement of co-occurring binge eating disorder in patients receiving topiramate for treatment of mood disorders. In addition, topiramate was associated with anorexia and weight loss in clinical trials with epilepsy patients. Also, topiramate has been demonstrated efficacy in pilot and controlled studies for binge eating disorder (BED) associated with obesity. Genetic studies will be important to elucidate the mechanism by which putative susceptibility variation in candidate genes influences in pharmacological improvement of binge eating disorder in obese patients treated with topiramate.

Connecting drug response with relevant functional DNA variants and differences in brain regions represents the ultimate goal for pharmacogenetic research playing an important role in advancing this understanding. The use of brain imaging combined with genetics can aid in understanding the pathophysiological mechanism of the disease. Additionally, brain imaging has the ability to bridge between preclinical research and human pharmacological studies.

This will be a naturalistic clinical study designed to analyze the effect of genetic variants and neurofunctional brain areas associated with food craving in patients with obesity and binge eating disorder responders to topiramate.

Hypothesis: The use of topiramate in obese subjects with binge eating disorder is associated with a differential gene variants and different activation brain areas in subjects that showed a reduction of food craving and weight lost.

DETAILED DESCRIPTION:
Obesity has been declared the number one illness of the 21st Century in industrialized countries, and is reaching epidemic proportions. Adoption, twin and family studies have reported that obesity has a strong heritable component and in particular, it has been suggested that BMI in adults is due to genetic influence rather than shared family environment. Binge eating in obese patients was escribed. Therefore, it has been proposed that binge eating disorder (BED) may contribute to obesity in some individuals. Subjects with BED are frequently obese. Conversely, BED is often observed in obese populations, especially the severely obese. Therefore, these findings suggest that BED is a major public health problem and a contributor to the obesity epidemic.

Evidence from twin studies suggests a significant contribution of genetic factor in binge eating. Interestingly, it was reported that relatives of patients with BED displayed a higher prevalence of obesity, particularly of severe obesity than relatives of probands without BED. Adoption and twin studies have consistently shown that, regardless of the population studied, genetic factors play an important role in determining the risk of developing binge eating.

Pharmacological studies reported that topiramate plays an important role in the treatment of binge eating disorder. It has been observed improvement of co-occurring binge eating disorder in patients receiving topiramate for treatment of mood disorder. In addition, topiramate was associated with anorexia and weight loss in clinical trials with epilepsy patients. Also, topiramate has been demonstrated efficacy in pilot and controlled studies for binge eating disorder (BED) associated with obesity. A paper review showed that topiramate weigtht loss was reported in 21 of 32 studies analyzed.

Recently, it was approved on 4/6/2012 the use of topiramate in combination with phentermine (QNEXA) in the Meeting of the Endocrinologic and Metabolic Drugs Advisory Committee of the Food and Drug Administration, as an adjunct to diet and exercise for weight management in patients with a body mass index (BMI) equal to or greater than 30 kilograms (kg) per square meter or a BMI equal to or greater than 27 kg per square meter if accompanied by weight-related co-morbidities.

Finally, animal studies have shown that stimulation of the lateral hypothalamus by glutamate and glutamate agonists, including kainite/AMPA agonists, causes an intense, rapid, dose-dependent increase in food intake.

Topiramate weight loss was reported in 21 of the 32 studies analysed and reached 5% reduction of the baseline weight prior treatment in 5 studies. Among the studies analyzed, a frequent finding was that the grater weight loss was associated with higher BMI at baseline. Also, diabetic patients were related with glycemic control and normalization of blood pressure in hypertensive subjects. Topiramate was generally well tolerated and serious adverse events were rare. Also, the use of topiramate was reported effective for weight reduction and improvement in glycemic control in obese subject with type 2 diabetes treated with metformin monotherapy.

Topiramate, which is approved for use in epilepsy and migraine prophylaxis, has multiple sites of action that might contribute to its neurostabilizing effects.

The mechanism of action of topiramate in BED is unknown. It may act as an appetite suppressant or satiety enhancer or somehow influence the reward system acting on appetite, and thereby reduce binge eating. Topiramate has not been shown to affect serotoninergic neurotransmission. Indeed, it has been shown to attenuate nicotine-induced increases in mesolimbic extracellular dopamine and norepinephrine, but not serotonin, release.

In addition, topiramate antagonizes glutamate receptors. Since glutamate and glutamate agonists rapidly elicit intense eating when injected into the lateral hypothalamus of rats, topiramate might reduce binge eating through glutamate antagonism. However, the mechanism of action of topiramate is unknown. Therefore, it is very important pharmacogenetic and neurofunctional brain studies that could help to elucidate the role of topiramate such as a new treatment for binge eating disorder associated with obesity in Mexican population.

Genetic studies will be important to elucidate the mechanism by which putative susceptibility variation in candidate genes influences in pharmacological improvement of binge eating disorder in obese patients treated with topiramate. DNA variants in coding and regulatory regions of genes will be both useful for systematic genome scans, for identifying genes associated with drug response, and for examining integrated systems of gene pathways as an important step on the route to functional genomics. Initiatives focused on identification of gene variants would greatly facilitate postgenomic research on the links between genes, brain, behavior, and treatment response.

Many drug targets (e.g., receptors, transporters, enzymes) that contribute to the pharmacodynamics of drug response are not only key players in the regulation of neurotransmitter systems but also directly or indirectly modify the development and plasticity of neural networks involved in drug effects. There is now considerable evidence that variability of epigenetic profiles of genes critical to neurocircuit development and function influences drug responses.

There are a number of different kinds of natural genetic variation that result in functional protein differences and affect drug responsiveness. The type of variation that is most prevalent in the genome and, arguably, the most relevant to common diseases and complex traits is represented by single nucleotide polymorphisms (SNPs).

There are many ways in which genetic variability, the differences in the sequence of specific genes, can lead to variability in drug responsiveness and it is likely that each of these mechanisms is involved in determining the effects for example in anticonvulsant drugs. Up to now, the focus of pharmacogenetic studies has been on "polymorphic drug metabolism". This methodology examines variations in the sequence of genes that code for drug-metabolizing enzymes. SNPs have been found to underlie variability in drug-metabolizing capacity and such variability is often documented as differences in drug and metabolite profiles between patients. It is likely that variation in genes coding for proteins involved in other pharmacokinetic processes, including drug absorption, distribution, and excretion, also help to determine individual differences in responsiveness although these mechanisms are not as well studied regarding genetic influences.

Another way in which genetic variation plays a role in drug responses depends upon polymorphisms in genes that code for proteins involved in drug targets or that mediate drug action. These differences in response apply both to therapeutic effects and adverse effects so that both efficacy and toxicity may be influenced by individual genetic variation. In the future, pharmacogenetic discoveries related to drugs will make individualization of therapy even more difficult in the sense that the genetic substrate that mediates efficacy may well differ from that mediates toxicity. As such, two different sets of genes and genotypes will need to be examined in order to match patients with the most appropriate treatment.

Differences in response apply both to therapeutic effects and adverse effects so that both efficacy and toxicity may be influenced by individual genetic variation.

In addition, compounds exist with mechanisms of action that either differ from standard drugs or are not yet fully characterized. These compounds and their mechanisms will lead eventually to the investigation of specific, possibly novel, genes in relation to drug responsiveness. Because behavioral traits are the most complex traits of all, response to psychopharmacological drugs, which modify behaviour traits, is likely to profit from this integration. Moreover, behavioural pharmacogenetics will make a major contribution to functional genomics.

Connecting drug response with relevant functional DNA variants and differences in brain regions represents the ultimate goal for pharmacogenetic research playing an important role in advancing this understanding. Brain imaging can provide valuable links in understanding the potential importance and clarifying the pathophysiological mechanisms that lie between associations of genetic variability and clinical response. Analysis of additional populations, such as Mexican population, is also necessary to achieve these goals. The use of brain imaging combined with genetics can aid in understanding the pathophysiological mechanism of the disease. Additionally, brain imaging has the ability to bridge between preclinical research and human pharmacological studies.

This study proposes the collection of samples which will result from this study will form the basis with which to identify the genes associated with neurofunctional brain areas involved in food craving in obese patients with BED treated with topiramate in Mexican population. The pharmacogenetic analysis in obese patients associated with BED will identify gene variants associated with the treatment efficacy to topiramate in Mexican population.

Objective The main objective of this study is to analyze the genetic variants and neurofunctional brain areas associated with food craving in obese patients with binge eating disorder responders to topiramate treatment.

Study design:

This will be a naturalistic clinical study designed to analyze the effect of genetic variants and neurofunctional brain areas associated with food craving in patients with obesity and binge eating disorder responders to topiramate.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of Eating Disorders Clinic with a diagnosis of Bulimia Nervosa, Eating Disorders Not Otherwise Specified 3 and 6 with Binge Eating Disorder according to research criteria in Diagnostic and Statistical of Mental Disorders, version IV revised, who started taking Topiramate.
2. Probands with diagnosis of obesity (BMI ≥30 kg/m2- 40 kg/m2).
3. Capable to give written informed consent.
4. Age of 18 to 50 years at screening.
5. Maternal and paternal grandparents of Mexican descent.
6. Probands without psychopharmacological treatment (including anticonvulsants) at least 4 weeks before inclusion.

Exclusion Criteria:

1. Subjects with alcohol or substance abuse or dependence.
2. Any psychiatric or medical disorder that requires inpatient treatment.
3. Psychosis or suicidal thoughts.
4. Abnormal blood chemistry.
5. Diabetes uncontrolled.
6. Unstable hypertension or difficult to control (criterion 7 of inclusion section).
7. Metabolic acidosis.
8. Narrow-angle glaucoma.
9. Unstable hypothyroidism or hyperthyroidism.
10. Unable or unwilling to give a blood sample.
11. Pace-makers or metal implants that would preclude the functional Magnetic Resonance Image scan.
12. Pregnant or lactating women at screening or positive blood pregnancy test.
13. Presence of any epileptic disorder.
14. Subjects unable or unlikely to follow the protocol procedures.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: This will be a single-center study that will seek to recruit 60 obese subjects with binge eating disorder who started taking Topiramate. Eligible male or female subjects, from or referred to, the Eating Disorder Clinic will be invited to participate in the study. Obesity will be defined as having a body mass index ≥ 30 kg/m2.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2013-06; Primary Completion 2013-12 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Treatment efficacy to topiramate in obese patients with binge eating disorder. | 6 weeks
  Topiramate will be initiated in all subjects at a 25 mg/day dose QD followed by a weekly increase of 25 mg/day and titrated until meaningful clinical response is obtained on binge episodes weekly frequency, binge/days weekly frequency. Meaningful clinical response is defined as a reduction to at least 50% on this parameter taking into account each individual's basal frequencies of binge and food craving. Maximum dose will be set at 400 mg/day (Arnone et al., 2005; McElroy et al., 2003; Shapira et al., 2000).

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz E Camarena, PhD, Principal Investigator — Instituto Nacional de Psiquiatria Dr. Ramon de la Fuente; Alejandro Caballero, M.D., Study Chair — Instituto Nacional de Psiquiatria Dr. Ramon de la Fuente; Juan J Cervantes, M.D., Study Chair — Instituto Nacional de Psiquiatria Dr. Ramon de la Fuente; Griselda Flores, M.D., Study Chair — Instituto Nacional de Psiquiatria Dr. Ramon de la Fuente; Sandra Hernandez, B,Sc., Study Chair — Instituto Nacional de Psiquiatria Dr. Ramon de la Fuente
Locations (1):
- Instituto Nacional de Psiquiatria Ramon de la Fuente Muñiz, México, D.f., Mexico